CLINICAL TRIAL: NCT03566615
Title: Does the Addition of a Cap Improve the Adenoma Detection Rate During Water Exchange Colonoscopy
Brief Title: Does the Cap Increase the Finding of Polyps When Water Exchange Colonoscopy is Used
Acronym: ASGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Felix W. Leung, Site PI and Director of Study, VA Greater Los Angeles Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: ASGE 2016 International Award
Record Dates: First submitted 2018-04-30; First posted 2018-06-25 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Colonoscopy; Polyp of Colon
Keywords: colonoscopy; adenoma detection rate; caps
MeSH Terms: conditions — Colonic Polyps; Cryopyrin-Associated Periodic Syndromes | interventions — Water

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water (Active Comparator): Residual air in the colon will be removed, water will be infused to guide insertion through an airless lumen. Infused water will be removed by suction, along with residual fecal debris, predominantly during insertion.
  Interventions: Other: water
- CAP-straight (Experimental): A straight transparent cap was fitted to the colonoscope per manufacturer instruction.Residual air in the colon will be removed, water will be infused to guide insertion through an airless lumen. Infused water will be removed by suction, along with residual fecal debris, predominantly during insertion.
  Interventions: Device: CAP-straight; Other: water
- CAP-daisy (Experimental): A daisy cap transparent cap was fitted to the colonoscope per manufacturer instruction.Residual air in the colon will be removed, water will be infused to guide insertion through an airless lumen. Infused water will be removed by suction, along with residual fecal debris, predominantly during insertion.
  Note:
  IRB Approval date for the use of Endocuff at St. Barbara Hospital, Iglesias (CA), Italy, was obtained on 3/8/2017.
  IRB Approval date for the use of Endocuff at Evergreen General Hospital, Taipei, Taiwan, was obtained on 3/18/2021.
  Interventions: Device: CAP-daisy; Other: water

INTERVENTIONS:
Device: CAP-straight — This study is to detect any differences in the detection rate of adenomas using straight caps that will be attached to the colonoscope and to compare it to the control method where no cap is used in the colonoscopy procedure.
  Arms: CAP-straight
Device: CAP-daisy — This study is to detect any differences in the detection rate of adenomas using daisy caps that will be attached to the colonoscope and to compare it to the control method where no cap is used in the colonoscopy procedure.
  Arms: CAP-daisy
Other: water — using water instead of traditional air insufflation to help insertion

SUMMARY:
This is a study to compare two different, but normally, used methods of colonoscopy in patients that require a routine or repeat colonoscopy. There will be three arms in this study: WE water control, water plus Cap-1, and water plus Cap-2. The patient will prepare himself/herself for the colonoscopy as per normal instructions and he/she will be given the information for the study at that time so that he/she can make a decision to participate in the study. The control method will use water instead of air inserted into the colon. The study method will use a new accessory, a cap that will fit onto the end of the colonoscope plus water during the procedure. This study will also confirm if using the cap method with water is a better way of detecting polyps in the colon and possibly cancer.

DETAILED DESCRIPTION:
This will be a multi-site, multi-national, unblinded investigators, prospective Random Control Trial (RCT). Randomization (WE, WE Cap-1, WE Cap-2) will be based on computer generated random numbers placed inside opaque sealed envelopes. The envelope (in pre-arranged order) will be opened to reveal the code when the colonoscopist is ready to insert the endoscope to begin the examination. This will be a comparison of two different methods with three arms (WE, WE Cap-1, WE Cap-2) to see which one is better at detecting adenomas.

Patients who are willing to participate will sign an informed consent before starting the colonoscopy procedure. Separate parallel randomization will be set up at each site, stratified by investigator and type of colonoscopy (screening or surveillance). Mode of sedation will include unsedated (China, US West Los Angeles VA), minimally sedated (Taiwan), on demand sedation (Italy, Czech Republic, US West Los Angeles VA), conscious sedation (US Sacramento VA and Palo Alto VA) or full sedation with propofol (Taiwan). Randomization (prepared by statistics consultant) will be carried out by the method of random permuted block design (based on computer generated random numbers) with variable block sizes of 3 and 6. Gender will be used as a stratification factor.

Control Method: One arm of the study will include sedated/unsedated colonoscopy with water (WE) as the control method. Residual air in the colon will be removed and water will be infused to guide insertion through an airless lumen. Infused water will be removed by suction, along with residual fecal debris, predominantly during insertion.

Study method: The other two arms entail the addition of a simple commercially available accessory to the colonoscopy device: Cap -1 (Disposable Distal Attachment) or Cap-2, fitted to the colonoscope per manufacturer instruction. The two arms include sedated/unsedated colonoscopy with either a Cap-1 plus water or Cap-2 plus water.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female 50-75 yrs of age.
2. Positive screening for Fecal Immunochemical Test (FIT) or Fecal Occult Blood Test (FOBT).
3. Subjects willing to undergo routine screening and surveillance colonoscopy.

Exclusion Criteria:

1. Patients who decline to provide informed consent.
2. Patients known to have colonic obstruction, inflammatory bowel disease, or active GI bleeding requiring interventions.
3. Patients know to have prior history of severe diverticulitis/diverticulosis.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1630 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 2 years
  The proportion of individuals undergoing a complete screening colonoscopy who have one or more adenomas, or polyps, detected.

SECONDARY OUTCOMES:
Cecal intubation | 2 hours: Data collected during colonoscopy procedure
  Visualization of ileocecal valve/appendix orifice and the medial wall of the cecum with colonoscope tip touching floor of cecum
Boston bowel preparation score | 2 hours: Data collected during colonoscopy procedure
  Three segments (Right, transverse, left colon), each with 0 to 3 (poor to excellent); total scores = sum (10 point scale)
Cecal intubation time | 2 hours: Data collected during colonoscopy procedure
  Total time from insertion into the anus to arrival in the cecum
Visual analogue scale (0=not satisfied, 10=very satisfied) | 2 hours: Data collected during colonoscopy procedure
  Patient satisfaction
Willing to repeat | 2 hours: Data collected during colonoscopy procedure
  Visual analogue scale (0=not willing, 10=willing)

CONTACTS AND LOCATIONS:
Overall Officials: Felix W Leung, MD, Principal Investigator — VA Greater Los Angeles Healthcare System
Locations (7):
- United States (2):
  - Sacramento VAMC, VA Northern California Healthcare System, Mather, California
  - Veterans Affairs Palo Alto Healthcare System, Palo Alto, California
- Xijing Hospital of Digestive Diseases, Xi'an, China
- St. Barbara Hospital, Iglesias, Italy
- Taiwan (3):
  - Dalin Tzu Chi General Hospital, Chiayi City
  - Hualien Tzu Chi Hospital, Hualien City
  - Evergreen General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No